CLINICAL TRIAL: NCT01790386
Title: Equivalency Study of the CORA(R) and TEG(R) 5000 Systems
Brief Title: Equivalency Study of the TEG and CORA Hemostasis Systems
Status: Completed | Type: Observational
Sponsor: Coramed Technologies LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Coramed 01-144
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Heart Disease; Focus is on Testing Performance of CORA Hemostasis System.
Keywords: hemostasis; thromboelastography; coagulation; TEG
MeSH Terms: conditions — Heart Diseases; Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical Patients Group: Patients undergoing cardiovascular surgery and cardiology procedures
- Reference Ranges Group: Healthy volunteer subjects for determination of normal hemostasis parameter results

SUMMARY:
This study is being performed to obtain data about the CORA system, a new device that is currently being tested and is not yet cleared for sale in the United State by the Food and Drug Administration (FDA). The purpose of the study is to validate the CORA system by comparing the results of this test to that of the standard of care device called the TEG system. Both systems evaluate hemostasis, a highly complex and interactive process involving many protein and cellular elements, especially platelets, occurring in a series of interrelated phases, which results in either normal hemostasis or a tendency toward bleeding or clotting complications.

DETAILED DESCRIPTION:
The study protocol specifies testing using multiple reagents which are similar for both the CORA and TEG systems. Tests are run on blood samples taken from patients undergoing cardiovascular surgery and cardiology procedures, at two times throughout the procedure. The tests may be performed at three different pairs of times: Pre-Operation and Post-Protamine, or During Operation (Post-Heparin) and ICU, or Pre-Operation and ICU. Patients are selected at random for determination of which pair of times will be used, as long as the number of patients for each of the three groups is approximately the same. Following the protocol defined in CLSI Standard EP09-A2, equivalence between the two systems will be demonstrated if the conclusions from the Standard Section 7, Interpreting Results and Comparing to Internal Performance Criteria, are found to be acceptable.

The study protocol also specifies the testing of blood samples from normal, health volunteer subjects for the purpose of determining CORA System Reference Ranges for all of the reagents used in the study. Reference ranges will be constructed following the guidelines specified in CLSI Standard C28-A3c.

All blood samples drawn for this study will use venous blood. Whole blood is not used for these studies; only citrated or heparinized samples are used. All samples are repeated twice (run in duplicate tests). Quality Controls are run on both instruments at a frequency specified by the manufacturers. Results obtained from this testing are not used to make treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over (both groups)
* Age, gender, ace and disease state documented (both groups)
* In good health (Reference Ranges group only)

Exclusion Criteria:

* Subjects/patients under the age of 18 (both groups)
* On medications affecting hemostasis (Reference Ranges group)
* Having conditions or undergoing treatments affecting hemostasis (Reference Ranges group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For surgical group, and consented patient 18 years of age or over, going through a heart surgical procedure.
  For Reference Ranges group, helathy subjects 18 years of age or over, not taking medications, having conditions or undergoing treatments that would affect blood hemostasis.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measurement of differences in TEG and CORA hemostasis parameters per patient | Parameter differences assessed at completion of patient surgery

SECONDARY OUTCOMES:
Measurement of test subjects' CORA Hemostasis Parameters | Hemostasis parameters measured at time of test for each subject
  Measurement of CORA hemostasis parameters for healthy volunteer subjects is necessary to establish Reference Ranges for product.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Medstar Health Research Institute - Washington Hospital Center, Washington D.C., District of Columbia
  - Sinai Center for Thrombosis Research, Sinai Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania